CLINICAL TRIAL: NCT04991025
Title: Phase 2 Trial of Neoadjuvant Nivolumab + Platinum-based Chemotherapy + Certolizumab in Patients With Resectable Stages II-III Lung Cancers
Brief Title: Adding Certolizumab to Chemotherapy + Nivolumab in People Who Have Lung Cancer That Can Be Treated With Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-152
Record Dates: First submitted 2021-07-27; First posted 2021-08-05 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer; Lung Cancer Stage II; Lung Cancer Stage III
Keywords: Untreated Lung Cancer; resectable lung cancer; operable lung cancer; Certolizumab; Memorial Sloan Kettering Cancer Center; 21-152
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Pemetrexed; Gemcitabine; Carboplatin; Certolizumab Pegol; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with resectable stage II-III lung cancers (Adenocarcinoma) (Experimental): This is a single arm phase II study of neoadjuvant platinum-based chemotherapy + nivolumab + certolizumab in participants with resectable stage II-III lung cancers. There will be separate adenocarcinoma and squamous cell carcinoma cohorts.
  Interventions: Drug: Cisplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Carboplatin; Drug: Certolizumab; Drug: Nivolumab
- Participants with resectable stage II-III lung cancers (squamous cell carcinoma) (Experimental): This is a single arm phase II study of neoadjuvant platinum-based chemotherapy + nivolumab + certolizumab in participants with resectable stage II-III lung cancers. There will be separate adenocarcinoma and squamous cell carcinoma cohorts.
  Interventions: Drug: Cisplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Carboplatin; Drug: Certolizumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Cisplatin — Participants with lung adenocarcinoma will receive standard of care neoadjuvant cisplatin 75mg/m2 + pemetrexed 500mg/m2 intravenously on day 1 of a 21 day cycle. Participants with squamous cell lung carcinoma will receive cisplatin 75mg/m2 IV on day 8 of a 21 day cycle + gemcitabine 1000mg/m2 IV days 1 and 8 of a 21 day cycle.
Drug: Pemetrexed — Participants with lung adenocarcinoma will receive standard of care neoadjuvant cisplatin 75mg/m2 + pemetrexed 500mg/m2 intravenously on day 1 of a 21 day cycle
Drug: Gemcitabine — Participants with squamous cell lung carcinoma will receive cisplatin 75mg/m2 IV on day 8 of a 21 day cycle + gemcitabine 1000mg/m2 IV days 1 and 8 of a 21 day cycle.
Drug: Carboplatin — Participants not eligible for cisplatin (per treating physician discretion) may receive carboplatin at AUC = 5 instead of cisplatin.
Drug: Certolizumab — Certolizumab 400mg subq will be administered in clinic within 1 hour before the start of chemotherapy on day 1 of a 21 day cycle.
Drug: Nivolumab — Participants with lung adenocarcinoma will receive standard of care neoadjuvant cisplatin 75mg/m2 + pemetrexed 500mg/m2 + nivolumab 360mg intravenously on day 1 of a 21 day cycle Participants with squamous cell lung carcinoma will receive cisplatin 75mg/m2 IV on day 8 of a 21 day cycle + gemcitabine 1000mg/m2 IV days 1 and 8 of 21 day cycle + nivolumab 360mg IV on day 1 of 21 day cycle.

SUMMARY:
The purpose of the study is to explore adding the study drug certolizumab to standard chemotherapy as it may reduce the inflammation caused by the cancer and make the chemotherapy more effective in shrinking the cancer. This study will examine whether adding certolizumab to the usual treatment approach is better than, the same as, or worse than the usual approach alone.

ELIGIBILITY:
Inclusion Criteria:

* Untreated stage II-III (AJCC 8th edition) non-small cell lung cancers with operable and resectable disease determined by a thoracic surgeon
* Histologic confirmation of disease at MSKCC
* Age 18 years or older
* Karnofsky Performance Status ≥ 70
* Adequate bone marrow, liver and renal function, as specified below:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9 /L
  * Lymphocyte count ≥0.5 x10^9/L (500/µL)
  * Hemoglobin ≥ 9 g/dL
  * Platelets ≥ 100 x 10^9 /L
  * Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) (except for patients with documented Gilbert's Syndrome)
  * AST and ALT ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 x upper limit of normal or creatinine clearance ≥ 60ml/min for patients with creatinine levels above institutional normal.
  * Serum albumin ≥25 g/L (2.5 g/dL)
  * For patients not receiving therapeutic anticoagulation: INR or aPTT ≤1.5 x ULN
  * For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Negative PPD test or interferon-gamma release assay (including but not limited to QuantiFERON-TB Gold)
* For women of child-bearing potential, negative pregnancy test within 14 days prior to starting treatment
* Men and women of childbearing age must be willing to use effective contraception while on treatment and for at least 5 months thereafter
* Presence of at least one site of measurable disease as defined by the Response Evaluation Criteria in Solid Tumors 1.1
* Ability to provide written, informed consent. Legally Authorized Representatives are permitted.
* Negative HIV test at screening, with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ³ 200/µL, and have an undetectable viral load
* Negative hepatitis B surface antigen (HBsAg) test at screening Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. Note: The HBV DNA test will be performed only for patients who have a negative HBsAg test and a positive total HBcAb test.
* Patient with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

* Presence of an FDA approved targeted therapy for patients with NSCLC harboring a genomic aberration for which an FDA-approved targeted therapy is indicated
* Hypersensitivity to platinum agents
* Prior use of TNF-α inhibitor
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment

Note: this exclusion criteria has the following excpetions:

* Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained.
* Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Topical steroids

  * Active or history of autoimmune disease or immune deficiency
  * Active or history of autoimmune disease or immune deficiency including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, psoriatic arthritis, antiphospholipid antibody syndrome Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis.

Note: This exclusion criteria has the following exceptions:

1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

   * Rash must cover < 10% of body surface area
   * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
   * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months

     * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted
     * Baseline hearing deficit (CTCAE version 4.0 grade 2 or higher)
     * Ongoing bacterial, viral, or antifungal infection requiring antimicrobial treatment with the exception of thrush
     * Active tuberculosis or untreated, latent tuberculosis Note: If a patient has signs, symptoms, or a history suggestive of active tuberculosis, evaluation by an infectious disease physician will be required and active tuberculosis ruled-out prior to enrollment.
     * Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, or cerebrovascular accident) within 3 months prior to initiation of study treatment, or unstable arrhythmia Note: Patients are ineligible if they have a history of myocardial infarction or
     * Unstable angina within the past 12 months
     * Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
     * Acute or chronic Hepatitis B or C infection
     * Known HIV infection requiring antiretroviral medications and those with AIDS
     * Active herpes zoster infection
     * Current treatment with anti-viral therapy for HBV
     * Non-healed infected skin ulcers
     * Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5mmol/L, calcium > 12mg/dL or corrected serum calcium > ULN)
     * Prior history of other malignancy with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, Stage I uterine cancer, localized prostate cancer, non-melanomatous skin cancer, ductal carcinoma or lobular carcinoma in situ of the breast
     * Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
     * Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment Note: Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
     * Prior allogeneic stem cell or solid organ transplantation
     * Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
     * Live, attenuated vaccines (e.g., FluMist) are prohibited within 4 weeks prior to initiation of study treatment, during treatment with nivolumab, and for 5 months after the last dose of nivolumab.
     * Treatment with investigational therapy within 28 days prior to initiation of study treatment
     * Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
     * Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
     * History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
     * Known hypersensitivity to Chinese hamster ovary cell products or to any component of the nivolumab formulation
     * Known allergy or hypersensitivity to any component of the Certolizumab pegol formulation
     * Known allergy or hypersensitivity to any component of the platinum-based chemotherapy formulations
     * Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of nivolumab, within 3 months after the final dose of Certolizumab pegol, and within 6 months after the final dose of carboplatin, cisplatin, pemetrexed or gemcitabine treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Participants complete pathologic response (CPR) | up to 2 years
  To evaluate the complete pathologic response (CPR) of participants with stage II-III lung cancers who receive treatment with neoadjuvant platinum-based chemotherapy + certolizumab pegol. Major pathologic response (MPR) is defined as 10% or less residual viable tumor after neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Paul Paik, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge Limited Protocol Activities, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org